CLINICAL TRIAL: NCT05536206
Title: Continuous and Wireless Vital Sign Monitoring in Patients at Home After Acute Medical Admission
Acronym: WARD-HOME
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Emilie Sigvardt, MD, Bispebjerg Hospital
Other Study IDs: H-20009132; WARD-HOME feasibility (Other: Bispebjerg Hospital)
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Vital Sign Monitoring; Clinical Deterioration; Disease Progression; Disease Attributes
MeSH Terms: conditions — Clinical Deterioration; Disease Progression; Disease Attributes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed patients: Adult patients (≥18 years) admitted with an acute medical disease and who are scheduled for discharge to their own homes within five days from inclusion.
  Interventions: Device: Wireless and continuously monitoring

INTERVENTIONS:
Device: Wireless and continuously monitoring — Included patients are monitored with WARD equipment during the last part of hospitalization and the first days after discharge with data transmitted in real time to personnel at the hospital. Monitoring will last for a maximum of 72 hours.

SUMMARY:
The current study aims to investigate the feasibility of transmitting continuous and wireless vital sign data in real time from patients home to the hospital in patients discharged after an acute medical hospitalization

DETAILED DESCRIPTION:
The healthcare system is challenged by an aging patient population with chronic diseases, and acute admissions must be housed in hospitals with fewer beds and less staff resources. This increases the need for earlier discharge and for treatment shifted to the patients' own home. Furthermore, the transition from the hospital to the home setting is one of potential hazard, due to the lack of observation and intervention possibilities.

This study aims to investigate the feasibility of wireless, continuous monitoring of patients in the days around discharge after an acute medical hospitalization, as well as occurrence of deviating vital signs i in the patients' own homes during the first days after discharge. Data will be transmitted continuously in real time from patient's homes to mobile applications for portable handheld devices such as healthcare personnel's smartphones.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) Admitted with an acute medical disease and scheduled for discharge to their own homes within five days from inclusion.

Exclusion Criteria:

* Allergy to plaster, plastic, or silicone.
* A pacemaker or Implantable Cardioverter Defibrillator (ICD) device.
* If the patient was deemed not able to open the front door when visited by the investigator.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with an acute medical disease at Bispebjerg Hospital and scheduled for discharge to their own homes within five days from inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Duration of data collection from the Lifetouch patch | Up to 72 hours of monitoring

SECONDARY OUTCOMES:
Duration of complete peripheral saturation data | Up to 72 hours of monitoring
Duration of complete blood pressure data | Up to 72 hours of monitoring
Cummulated duration of desaturation | Up to 72 hours of monitoring
  Peripheral saturation below 88% and 85%
Number of events with SpO2 < 88% in at least 10 consecutive minutes | Up to 72 hours of monitoring
Number of events with SpO2 < 85% in at least 5 consecutive minutes | Up to 72 hours of monitoring
Number of deviating vital parameters in accordance to defined microevents | Up to 72 hours of monitoring

OTHER OUTCOMES:
Re-admission and cause of re-admission within 30-days | 30-days follow up
User experiences (patient and personnel) | Within 72 hours of monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Sigvardt, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: No